CLINICAL TRIAL: NCT03292718
Title: Innovative Approach for Self-management and Social Welfare of Cystic Fibrosis Patients in Europe: Development, Validation and Implementation of a Telematics Tool. WP6.2: Impact Assessment Through a European Multicentre Clinical Trial: Validation of MyCyFAPP as a Portable System for Self-management in Children With CF
Brief Title: Clinical Trial to Assess Influence of MyCyFAPP Use on GI Related QOL in Children With Cystic Fibrosis
Acronym: MyCyFAPP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: Hospital Universitario La Fe (Other); European Commission (Other)
Responsible Party: Principal Investigator, Mieke Boon, MD PhD, Mieke Boon, Universitaire Ziekenhuizen KU Leuven
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: s60787
Record Dates: First submitted 2017-09-20; First posted 2017-09-25 (Actual); Last update posted 2017-09-25 (Actual); Status verified 2017-09

CONDITIONS: Cystic Fibrosis in Children
Keywords: PERT; mobile application

STUDY DESIGN:
Intervention Model Description: Single group, open label, with intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- use of MyCyFAPP (Experimental): use of MyCyFAPP during 6 months
  Interventions: Device: MyCyFAPP

INTERVENTIONS:
Device: MyCyFAPP — use of the MycyFAPP with all its features during 6 months

SUMMARY:
Interventional trial to study the influence of the use of MyCyFAPP (mobile application) on the gastro-intestinal related quality of life.

This mobile APP has been developed during previous workpackages of the Horizon2020 Project and contains several modules:

* mathematical prediction model to calculate the needed dose for pancreatic enzyme replacement therapy
* educational games and other educational material
* communication with doctor/dietician through professional webtool
* diary to register symptoms and data on nutrition.

The app will be introduced and used during 6 months. Primary outcome parameter will be change in modified PedsQL GI after 3 months. PedsQL GI is an existing questionnaire that evaluates gastro-intestinal related quality of life in children. We validated it for use in cystic fibrosis in a previous observational study.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of CF as evidenced by one or more clinical feature consistent with the CF phenotype or positive CF newborn screen AND one or more of the following criteria:

   1. A documented sweat chloride ≥ 60 mEq/L by quantitative pilocarpine iontophoresis (QPIT)
   2. A documented genotype with two disease-causing mutations in the CFTR gene
2. Having pancreatic insufficiency (stool elastase < 200 mcg/g stool) and using PERT
3. Age ≥ 24 months and < 18 years at screening visit
4. Informed consent by parent or legal guardian; assent for children from age 12 years on

6. Inclusion visit coincides with scheduled routine clinic visit 7. Ability and willingness to comply with APP use and evaluations at time of routine clinic visits as judged by the site investigator 8. Availability of wifi connection at home so that connection to the internet is feasible at home at least weekly.

Exclusion Criteria:

1. Acute infection associated with decreased appetite or fever at time of run-in visit
2. Acute abdominal pain necessitating an intervention at time of run-in visit
3. Physical findings that would compromise the safety of the participant or the quality of the study data as determined by site investigator
4. Investigational drug use within 30 days prior to run-in visit
5. Started with CFTR modulator treatment less than 3 months before start of run-in visit
6. Inability to use the APP due to patient specific factors such as language or learning difficulties

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 200 (Estimated)
Dates: Start 2017-10 (Estimated); Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
change in Modified PedsQL GI | 3 months
  Modified PedsQL GI will be assessed at month 0 and month 3 by applying questionnaires to children and their parents

SECONDARY OUTCOMES:
change in CFQ-R | 3 months and 6 months
  CFQ-R will be assessed by questionnaires
change in VAS | 3 months and 6 months
  VAS will be assessed by questionnaires
change in Modified PedsQL GI | 6 months
  Modified PedsQL GI will be assessed at month 0 and month 6 by applying questionnaires to children and their parents
change in lung function | 3 and 6 months
  spirometry will be performed

REFERENCES:
- See also: Related Info — http://www.mycyfapp.eu/en/